CLINICAL TRIAL: NCT07345117
Title: From Research to Clinical Practice: Implementation of an Internet-based Transdiagnostic Treatment Program for Emotional Disorders in Primary Care (TREAT-ED)
Brief Title: Cost-effectiveness and Implementation of a Transdiagnostic Internet-based Intervention for Emotional Disorders in Community Care.
Acronym: TREAT-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital Universitari Mutua Terrassa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTon-Terrassa
Record Dates: First submitted 2025-09-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Emotional Disorders; Depression Anxiety Disorder; Depression Disorders; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdiagnostic intervention protocol (Experimental): Internet-based psychological intervention (UJI online transdiagnostic protocol). This protocol, based on the transdiagnostic perspective, offers the possibility of applying a single psychological treatment for different emotional disorders by proposing that these disorders share a common vulnerability which, associated with certain stress factors, gives rise to different manifestations of this vulnerability (depression and various anxiety disorders).
  Interventions: Behavioral: Internet-based psychological intervention
- Treatment as usual (TAU) (Active Comparator): Standard treatment administered at participating health centers.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Internet-based psychological intervention — This protocol consists of a set of techniques that have proven effective in improving the lives of people with emotional disorders and is designed to be applied via the Internet. Its objective is to teach strategies that improve the ability to regulate emotions in a more adaptive way.
  It includes the following core therapeutic components, aimed primarily at regulating negative affect: a) emotional awareness focused on the present moment and acceptance, b) cognitive flexibility, c) emotional and behavioral avoidance, and d) exposure to emotional experiences (interoceptive and situational). In addition, the protocol also includes traditional evidence-based components for the treatment of emotional disorders, such as psychoeducation, motivation for change, and relapse prevention. Finally, it also includes a specific component for regulating positive affect, with the aim of promoting psychological strengths and improving well-being.
  Other Names: UJI online transdiagnostic protocol
  Arms: Transdiagnostic intervention protocol
Behavioral: Treatment as usual (TAU) — TAU may include pharmacological treatment (antidepressants and/or anxiolytics), psychological treatments (case management, group therapy, empathic listening, and counseling and advice), mental health nursing follow-up with psychosocial interventions, or a combination thereof. Participants in TAU and receiving treatment outside the center will be excluded from the study. The specific treatment received by each patient will be recorded. After the study, TAU participants will be given access to online treatment.
  Arms: Treatment as usual (TAU)

SUMMARY:
Emotional disorders (ED) are one of the leading causes of disability. They are highly prevalent and have an impact on quality of life. Addressing them places an overload on the National Health System (NHS), generating waiting lists and limiting appropriate care. The need for cost-effective solutions has led to the consideration of the transdiagnostic approach and the use of digital solutions. Both perspectives have demonstrated efficacy in a large number of randomized clinical trials. As a result, investment in digital health interventions is on the rise to improve access to care in overburdened healthcare systems. However, their integration and implementation in health systems remains limited. Implementation Science emerges to facilitate the integration of interventions into clinical practice through specific strategies that overcome barriers and optimize their sustainability. The objective of this project is to examine the effectiveness, economic costs and feasibility of implementing an online psychological treatment program for emotional disorders in mental health services. The Mutua and UJI teams have already carried out the transfer of the online program. In order to facilitate the adoption and sustainability of this program and that it can be used by mental health professionals in daily practice, a hybrid design 1 study will be carried out in which not only the efficacy but also the possibility of adoption and the analysis of economic costs in comparison with the usual treatment will be evaluated.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines mental health as "a state of well-being in which every individual realizes his or her potential, can cope with the stresses of life, can work productively and fruitfully, and is able to make a contribution to his or her community." Many people do not achieve this state of well-being, or even if they do, they lose it at some point in their lives. When this happens, it can take the form of a mental disorder, the most prevalent being depressive and anxiety disorders, which affect around 6% of the population in Spain, causing a major impact on their social, work, and personal lives. In the wake of the COVID pandemic, there has been greater awareness in society of the importance of mental health.

However, despite this and despite the availability of effective pharmacological and psychological treatments that can significantly alleviate the symptoms of many mental disorders, health systems are not responding adequately to people with mental disorders. A study exploring mental health care in 84 countries, including Spain (Moitra et al., 2022), found that only 23% of people with depression in high-income countries and 3% in middle-income countries received minimally adequate treatment for their problem. This indicates that the problem goes beyond a health issue; it is a social and ethical problem, since without adequate treatment, many mental disorders have very negative consequences that significantly reduce well-being, satisfaction, and quality of life and cause social inequalities.

Possible solutions include increasing the number of professionals and organizing the provision of services more efficiently, from prevention to specialized care, including primary care. In this regard, there is a very solid line of research that has shown that online psychological treatments are as effective as face-to-face treatments for people with moderate depression and anxiety disorders. This project is part of the objective of optimizing mental health services by incorporating an online treatment program in order to increase citizens' access to effective psychological treatments.

The researchers involved in this application form a team that combines healthcare work with scientific work in order to implement an online transdiagnostic treatment program, going beyond individual face-to-face therapy, increasing diversity in the ways psychotherapy is administered, being flexible, and expanding the range of services offered. The team at the Universitat Jaume I (UJI) has developed and validated the "UJI online transdiagnostic protocol" in rigorous clinical trials and with the collaboration of affected individuals (user-centered design), which is effective in the short and long term for depression and anxiety. Over the past year, the UJI team and the Mutua Terrassa team, through a transfer agreement, have integrated the program into Mutua's technology platform. This application aims to promote the adoption and sustainability of this program as an additional alternative available to mental health professionals at the two mental health centers run by Mutua Terrassa, which serve a population of more than 200,000 inhabitants.

The idea is to offer this program to people with moderate depression and/or anxiety so that professionals can intensify face-to-face care for other patients with more serious conditions. A clinical trial will be conducted to compare the effectiveness and costs of the online program with the usual treatment received by patients. In addition, the opinions of professionals and patients about the program will be evaluated, and the barriers and facilitators of incorporating the online program into services will be analyzed. The results will indicate the usefulness of this alternative. If the results are positive, an affordable, evidence-based alternative will be available that will increase the scope and scalability of treatments, which will be more integrated into people's daily lives, expanding the settings in which interventions are provided, with the acceptance of those involved. The project's actions include a plan to disseminate the results to society through social media networks belonging to both the UJI and Mutua; the organization of a specific conference on the project's results for primary care and specialist professionals at Mutua and another conference for patient and user associations; and holding meetings with managers who can make decisions about the sustainability of the program and its adoption in other services (General Directorate of Mental Health of the Valencian Community, management, health, and executive boards of Catsalut).

ELIGIBILITY:
Patient Inclusion Criteria:

* Over 18 years of age.
* Meet the diagnostic criteria for an anxiety or depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Understand and read Spanish or Catalan.
* Have access to the Internet and an email address
* Give informed consent.

Patient Exclusion Criteria:

* Diagnosis of schizophrenia, bipolar disorder, or alcohol or substance dependence.
* High risk of suicide.
* Presence of a medical condition that prevents psychological treatment.
* Receiving other psychological treatment (other than TAU or the online program) during the study.
* For participants in the online treatment condition with pharmacological treatment, this must be stabilized (doses cannot be changed or increased during the study, only reduced).

Inclusion Criteria for mental health Professionals:

* They work at centers participating in the study.
* They agree to participate in the study.
* They sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Level of effectiveness of the intervention in reducing depressive symptoms using the Overall Depression Severity and Impairment Scale (ODSIS) | Baseline, at the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Scores equal to or greater than 5 discriminate patients with clinical depressive symptoms.
Level of effectiveness of the intervention in reducing anxiety symptoms using the Overall Anxiety Severity and Impairment Scale (OASIS) | Baseline, at the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Scores equal to or greater than 7 discriminate patients with symptoms of clinical anxiety.
Level of effectiveness of the intervention in improving positive and negative affect using the Positive and Negative Affect Scale (PANAS) | Baseline, at the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  2 subscales: Negative and Positive Affect. Higher scores in each subscale indicates more neuroticism and positive affect, respectively.
Level of effectiveness of the intervention in improving quality of life using the EuroQoL-5D-3L | Baseline, at the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  This questionnaire describes health status in terms of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) according to five levels of severity. The experimental group will experience a more substantial improvement in quality of life compared to the TAU group, as evidenced by superior outcomes on the European Quality of Life 5D (EUROQOL).

SECONDARY OUTCOMES:
Level of acceptability of the intervention using the System Usability Scale (SUS) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Cut-off: a score of 68 and higher is considered acceptable usability.
Level of acceptability of the intervention using the Acceptability of Intervention Measure (AIM) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Cut-off scores for interpretation are not yet available; however, higher scores indicate greater acceptability.
Level of acceptability of the intervention using the Client Satisfaction Questionnaire adapted to Internet-based interventions (CSQ-I). | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Cut-off scores for interpretation are not yet available; however, higher scores indicate greater client satisfaction and acceptability.
Level of feasibility of the intervention using the Feasibility of Intervention Measure (FIM) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Cut-off scores for interpretation are not yet available; however, higher scores indicate greater feasibility.
Level of feasibility of the intervention using passive data collected by the platform. | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Program usage metrics (module completion, dropout, and frequency of use).
Level of appropriateness of the intervention using the Intervention Appropriateness Measure (IAM) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Cut-off scores for interpretation are not yet available; however, higher scores indicate greater appropriateness.
Barriers and facilitators to intervention implementation measured quantitatively with the Pragmatic Context Assessment Tool (pCAT) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
Barriers and facilitators to intervention implementation measured qualitatively with semi-structured interviews and focus groups | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
  Following the Consensual Qualitative Research (CQR) guidelines
Cost analysis - Initial technology investment costs | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
Cost analysis - Direct costs using the ICT-P adult questionnaire | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.
Cost analysis - Indirect costs using the Productivity Costs Questionnaire (iPCQ) | At the end of the intervention and follow-up at 3, 6, 9 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Azucena Garcia-Palacios, Psychology, Study Director — Universitat Jaume I
Locations (1):
- Laboratorio de Psicología y Tecnología (LabPsiTec), Castellon, Castellon, Spain

REFERENCES:
- [Background] Gonzalez-Robles A, Suso-Ribera C, Diaz-Garcia A, Garcia-Palacios A, Castilla D, Botella C. Predicting response to transdiagnostic iCBT for emotional disorders from patient and therapist involvement. Internet Interv. 2021 Jun 20;25:100420. doi: 10.1016/j.invent.2021.100420. eCollection 2021 Sep. PMID 34401379
- [Background] Gonzalez-Robles A, Roca P, Diaz-Garcia A, Garcia-Palacios A, Botella C. Long-term Effectiveness and Predictors of Transdiagnostic Internet-Delivered Cognitive Behavioral Therapy for Emotional Disorders in Specialized Care: Secondary Analysis of a Randomized Controlled Trial. JMIR Ment Health. 2022 Oct 31;9(10):e40268. doi: 10.2196/40268. PMID 36315227
- [Background] Diaz-Garcia A, Gonzalez-Robles A, Garcia-Palacios A, Fernandez-Alvarez J, Castilla D, Breton JM, Banos RM, Quero S, Botella C. Negative and Positive Affect Regulation in a Transdiagnostic Internet-Based Protocol for Emotional Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Feb 1;23(2):e21335. doi: 10.2196/21335. PMID 33522977
- [Background] Gonzalez-Robles A, Diaz-Garcia A, Garcia-Palacios A, Roca P, Ramos-Quiroga JA, Botella C. Effectiveness of a Transdiagnostic Guided Internet-Delivered Protocol for Emotional Disorders Versus Treatment as Usual in Specialized Care: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 7;22(7):e18220. doi: 10.2196/18220. PMID 32673226
- See also: Mutua Terrassa website — https://www.mutuaterrassa.com/es/home
- See also: LabPsiTec website — https://www.labpsitec.uji.es/